CLINICAL TRIAL: NCT01765790
Title: A Phase 1 Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Anti-MIF Antibody in Subjects With Malignant Solid Tumors
Brief Title: Phase 1 Study of Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 391101; 2013-002870-31 (EudraCT Number)
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Adenocarcinoma of the Colon or Rectum; Malignant Solid Tumors
MeSH Terms: conditions — Colonic Neoplasms | interventions — Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Malignant Solid Tumor (Arm 1) (Experimental): Dose Escalation Phase- Standard dose escalation of anti-MIF antibody in 5 dose groups of 3-6 participants each according to 3+3 design: 1. Dose escalation will be performed after safety data review, following completion of dosing of each cohort. -> 2. Safety data review. If dose escalation permissible -> 3. Next dose group -> 4. Safety data review, etc.
  Dose Expansion Phase- Enrollment of up to 6 participants to receive anti-MIF antibody (at the maximum tolerated dose or lower) in order to gain further experience with the investigational product at a specific dose level(s).
  Interventions: Biological: Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody
- Metastatic Adenocarcinoma of the Colon or Rectum (Arm 2) (Experimental): Dose Escalation Phase- Standard dose escalation of anti-MIF antibody in 3 dose groups of 3-6 participants each according to 3+3 design: 1. Dose escalation will be performed after safety data review, following completion of dosing of each cohort. -> 2. Safety data review. If dose escalation permissible -> 3. Next dose group -> 4. Safety data review, etc.
  Dose Expansion Phase- Enrollment of up to 6 participants to receive anti-MIF antibody (at the maximum tolerated dose or lower) in order to gain further experience with the investigational product at a specific dose level(s).
  Interventions: Biological: Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody

INTERVENTIONS:
Biological: Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody — * Dosing every 2 weeks
  * Intravenous injection
  Arms: Malignant Solid Tumor (Arm 1)
Biological: Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody — * Dosing weekly
  * Intravenous injection
  Arms: Metastatic Adenocarcinoma of the Colon or Rectum (Arm 2)

SUMMARY:
The purpose of the study is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of anti-MIF antibody in subjects with malignant solid tumors (Arm 1) and in subjects with metastatic adenocarcinoma of the colon or rectum (Arm 2).

ELIGIBILITY:
Main Inclusion Criteria:

* Males and females 18 years of age and older at the time of screening
* Anticipated life expectancy > 3 months at the time of screening
* Arm 1 only: Histologically confirmed malignant solid tumor which is refractory to or has failed standard treatments, or participant is not considered medically suitable to receive standard of care treatment or refuses standard of care treatment
* Arm 2 only: Histologically or cytologically confirmed diagnosis of metastatic adenocarcinoma of the colon or rectum which is refractory to or has failed standard treatments, or participant is not considered medically suitable to receive standard of care treatment or refuses standard of care treatment
* Measurable or evaluable disease (as defined in the study protocol)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate hematological function (as defined in the study protocol)
* Adequate renal function (as defined in the study protocol)
* Adequate liver function (as defined in the study protocol)
* Adequate venous access
* Arm 2 only: At least 1 tumor that is amenable to biopsy, as determined by the investigator, and participant must be willing to undergo a biopsy prior to and at least once following anti-macrophage migration inhibitory factor (anti-MIF) antibody treatment
* For women of childbearing potential, the participant must have a negative pregnancy test at screening and must agree to employ 2 forms of adequate contraceptive measures
* For males, participants must agree to use adequate contraceptive measures including at least 1 barrier method, and abstain from sperm donation throughout the course of the study and for at least 90 days after the last administration of investigational product.
* Participant is willing and able to comply with the requirements of the protocol

Main Exclusion Criteria:

* Known brain tumors or Central nervous system (CNS) metastases
* Myocardial infarction within 6 months of anti-MIF antibody administration, congestive heart failure (New York Heart Association Class III or Class IV), unstable angina, unstable cardiac arrhythmia requiring medication, or risk factors for polymorphic ventricular tachycardia
* Uncontrolled hypertension
* Left ventricular ejection fraction (LVEF) <40%, as determined by screening echocardiogram (echocardiogram results obtained within 90 days prior to screening are acceptable)
* QT/QTc interval >450 msec, as determined by screening electrocardiogram (ECG)
* Antitumor therapy (chemotherapy, radiotherapy, antibody therapy, molecular targeted therapy, retinoid therapy, or hormonal therapy) within 4 weeks prior to administration of the investigational product (IP) (6 weeks for nitrosoureas and mitomycin C). Any previous treatment-related toxicities must have recovered to Grade ≤ 1 (graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03). Prior and concurrent use of hormone deprivation therapies for hormone-refractory prostate cancer or breast cancer are permitted.
* Major surgery within 4 weeks prior to IP administration
* Active joint inflammation or history of inflammatory arthritis or other immune disorder involving the joints
* Active infection requiring IV antibiotics within 2 weeks prior to screening
* Known history of hepatitis B virus (HBV), hepatitis C virus (HCV), or active tuberculosis. Known history of human immunodeficiency virus (HIV) type 1/2 or other immunodeficiency disease.
* Participant has received a live vaccine within 4 weeks prior to screening
* Known hypersensitivity to any component of recombinant protein production by Chinese Hamster Ovary (CHO) cells
* Participant has been exposed to an investigational product (IP) or investigational device in another clinical study within 4 weeks prior to IP administration, or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
* Participant is nursing or intends to begin nursing during the course of the study
* Any disorder or disease, or clinically significant abnormality on laboratory or other clinical test(s), that in medical judgment may impede the participant's participation in the study, pose increased risk to the participant, or confound the results of the study
* Participant is a family member or employee of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-06-14 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing serious adverse events (SAEs) and/or adverse events (AEs) regardless of causality | 14 months

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters | 28 days
  Maximum concentration (Cmax), minimum concentration (Cmin), area under the concentration vs time curve (AUC), half-life [t½], clearance (CL), mean residence time (MRT) and volume of distribution at steady state (VDss)
Tumor response | 14 months
Levels of free active MIF and free total MIF in plasma and tumor tissue (where applicable) | 14 months
Change in levels of tumor-associated biomarkers, if applicable based on cancer type, following treatment with anti-MIF antibody | 14 months
Number of serious adverse events (SAEs) and/or adverse events (AEs), regardless of causality | 14 Months
Number of participants experiencing related serious adverse events (SAEs) and/or adverse events (AEs) | 14 months
Number of related serious adverse events (SAEs) and/or adverse events (AEs) | 14 months
Number of dose limiting toxicities (DLTs) | 14 months
Number of participants experiencing dose limiting toxicity (DLT) | 14 months
Number of participants who develop binding and/or neutralizing anti-anti-macrophage migration inhibitory factor (anti-MIF) antibodies following treatment with anti-MIF | 14 months
Anti-MIF antibody in tumor tissues, bound and/or unbound to active MIF (where applicable) | 14 Months
Levels of other potential biomarkers in tumor tissue (where applicable) | 14 Months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (4):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Florida Cancer Specialists / Sarah Cannon Research Institute, Sarasota, Florida
  - Department of Investigator Cancer Therapeutics, University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center (CTRC), The University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mahalingam D, Patel MR, Sachdev JC, Hart LL, Halama N, Ramanathan RK, Sarantopoulos J, Volkel D, Youssef A, de Jong FA, Tsimberidou AM. Phase I study of imalumab (BAX69), a fully human recombinant antioxidized macrophage migration inhibitory factor antibody in advanced solid tumours. Br J Clin Pharmacol. 2020 Sep;86(9):1836-1848. doi: 10.1111/bcp.14289. Epub 2020 Apr 12. PMID 32207164